CLINICAL TRIAL: NCT00122460
Title: Cetuximab in Combination With Cisplatin or Carboplatin and 5-Fluorouracil in the First Line Treatment of Subjects With Recurrent and/or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Cetuximab (Erbitux) in Combination With Cisplatin or Carboplatin and 5-Fluorouracil in the First Line Treatment of Subjects With Recurrent and/or Metastatic Squamous Cell Carcinoma of the Head and Neck (EXTREME)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 62202-002
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Results first posted 2011-09-30 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cetuximab; Platinum; Cisplatin; Carboplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cetuximab Plus Chemotherapy (Experimental)
  Interventions: Drug: Cetuximab + Platinum (Cisplatin or Carboplatin) + 5Fluorouracil (5-FU)
- Chemotherapy alone (Active Comparator)
  Interventions: Drug: Platinum (Cisplatin or Carboplatin) + 5-FU

INTERVENTIONS:
Drug: Cetuximab + Platinum (Cisplatin or Carboplatin) + 5Fluorouracil (5-FU) — Subjects in will receive initial dose of 400 mg/m^2 cetuximab (over 2 hours) followed by weekly doses of 250 mg/m^2 (over 1 hour). All doses will be given by intravenous (IV) infusion. Subjects will receive either Cisplatin (100 mg/m^2 on day 1) + 5-FU (1000 mg/m^2 continuous IV from day 1 to day 4) every 3 weeks or Carboplatin (Area under the curve (AUC) 5 IV on day 1) + 5-FU (1000 mg/m^2 continuous IV from day 1 to day 4) every 3 weeks
  Arms: Cetuximab Plus Chemotherapy
Drug: Platinum (Cisplatin or Carboplatin) + 5-FU — All doses will be given by IV infusion. Subjects will receive either Cisplatin (100 mg/m^2 on day 1) + 5-FU (1000 mg/m^2 continuous IV from day 1 to day 4) every 3 weeks or Carboplatin (AUC 5 IV on day 1) + 5-FU (1000 mg/m^2 continuous IV from day 1 to day 4) every 3 weeks
  Arms: Chemotherapy alone

SUMMARY:
The purpose of this trial is to investigate the efficacy of cetuximab in combination with chemotherapy in comparison to chemotherapy alone in patients with recurrent or metastatic head and neck cancer. Overall survival will be taken as the primary measure of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of squamous cell carcinoma of the head and neck (SCCHN)
* Recurrent and/or metastatic SCCHN, not suitable for local therapy

Exclusion Criteria:

* Prior systemic chemotherapy, except if given as part of a multimodal treatment for locally advanced disease which was completed more than 6 months prior to study entry
* Surgery (excluding prior diagnostic biopsy), or irradiation within 4 weeks before study entry
* Nasopharyngeal carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2004-12; Primary Completion 2007-03 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (70):
- Austria (2):
  - Research Site, Innsbruck
  - Research Site, Vienna
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Ghent
- Czechia (2):
  - Research Site, České Budějovice
  - Research Site, Prague
- France (12):
  - Research Site, Caen
  - Research Site, Dijon
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nantes-Saint Herblain
  - Research Site, Nice
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Tours
  - Research Site, Vandœuvre-lès-Nancy
- Germany (7):
  - Research Site, Berlin
  - Research Site, Essen
  - Research Site, Frankfurt on the Main
  - Research Site, Hamburg
  - Research Site, Munich
  - Research Site, Oldenburg
  - Research Site, Stuttgart
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Kecskemét
  - Research Site, Nyíregyháza
- Italy (6):
  - Research Site, Cuneo
  - Research Site, Genoa
  - Research Site, Milan
  - Research Site, Monserrato
  - Research Site, Naples
  - Research Site, Rome
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Nijmegen
- Poland (3):
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Warsaw
- Portugal (2):
  - Research Site, Lisbon
  - Research Site, Porto
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Slovakia (2):
  - Research Site, Bratislava
  - Research Site, Košice
- Spain (8):
  - Research Site, Barcelona
  - Research Site, Donostia / San Sebastian
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Santander
  - Research Site, Seville
  - Research Site, Valencia
- Sweden (3):
  - Research Site, Lind
  - Research Site, Örebo
  - Research Site, Umeå
- Switzerland (3):
  - Research Site, Geneva
  - Research Site, Thun
  - Research Site, Zurich
- Ukraine (4):
  - Research Site, Donetsk
  - Research Site, Kharkiv
  - Research Site, Kiev
  - Research Site, Sumy
- United Kingdom (5):
  - Research Site, Chelmsford
  - Research Site, Edinburgh
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Nottingham

REFERENCES:
- [Result] Vermorken JB, Mesia R, Rivera F, Remenar E, Kawecki A, Rottey S, Erfan J, Zabolotnyy D, Kienzer HR, Cupissol D, Peyrade F, Benasso M, Vynnychenko I, De Raucourt D, Bokemeyer C, Schueler A, Amellal N, Hitt R. Platinum-based chemotherapy plus cetuximab in head and neck cancer. N Engl J Med. 2008 Sep 11;359(11):1116-27. doi: 10.1056/NEJMoa0802656. PMID 18784101
- [Result] Mesia R, Rivera F, Kawecki A, Rottey S, Hitt R, Kienzer H, Cupissol D, De Raucourt D, Benasso M, Koralewski P, Delord JP, Bokemeyer C, Curran D, Gross A, Vermorken JB. Quality of life of patients receiving platinum-based chemotherapy plus cetuximab first line for recurrent and/or metastatic squamous cell carcinoma of the head and neck. Ann Oncol. 2010 Oct;21(10):1967-1973. doi: 10.1093/annonc/mdq077. Epub 2010 Mar 24. PMID 20335368
- [Derived] Hecht M, Hahn D, Wolber P, Hautmann MG, Reichert D, Weniger S, Belka C, Bergmann T, Gohler T, Welslau M, Grosse-Thie C, Guntinas-Lichius O, von der Grun J, Balermpas P, Orlowski K, Messinger D, Stenzel KG, Fietkau R. Treatment response lowers tumor symptom burden in recurrent and/or metastatic head and neck cancer. BMC Cancer. 2020 Sep 29;20(1):933. doi: 10.1186/s12885-020-07440-w. PMID 32993574
- [Derived] Licitra L, Storkel S, Kerr KM, Van Cutsem E, Pirker R, Hirsch FR, Vermorken JB, von Heydebreck A, Esser R, Celik I, Ciardiello F. Predictive value of epidermal growth factor receptor expression for first-line chemotherapy plus cetuximab in patients with head and neck and colorectal cancer: analysis of data from the EXTREME and CRYSTAL studies. Eur J Cancer. 2013 Apr;49(6):1161-8. doi: 10.1016/j.ejca.2012.11.018. Epub 2012 Dec 19. PMID 23265711

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last subject(informed consent): 14Dec 2004/28 Dec2005. Clinical cut-off: 12 Mar 2007. 80 centers in Europe: Austria (3), Belgium (5), Czech Republic (2), France (12),Germany (8), Hungary (4), Italy (5), Netherlands (4), Poland (5), Portugal (3), Russia (4), Slovakia (2), Spain (9), Sweden (3), Switzerland (3), UK (4), and Ukraine (4).
Pre-assignment Details: 477 subjects screened. 41 ineligible for treatment at end of screening (inclusion/exclusion criteria not fulfilled (30),death (3),consent withdrawal(3), symptomatic deterioration(2),non-compliance with timelines(1),refusal to continue study procedures (1), missing (1).436 eligible for treatment; however 6 of the ineligible patients were randomized
Groups:
- Cetuximab Plus Chemotherapy: Subjects in will receive initial dose of 400 mg/m^2 cetuximab (over 2 hours) followed by weekly doses of 250 mg/m^2 (over 1 hour). All doses will be given by intravenous (IV) infusion. Subjects will receive either Cisplatin (100 mg/m^2 on day 1) + 5-FU (1000 mg/m^2 continuous IV from day 1 to day 4) every 3 weeks or Carboplatin (Area under the curve (AUC) 5 IV on day 1) + 5-FU (1000 mg/m^2 continuous IV from day 1 to day 4) every 3 weeks.
- Chemotherapy Alone: All doses will be given by IV infusion. Subjects will receive either Cisplatin (100 mg/m^2 on day 1) + 5-FU (1000 mg/m^2 continuous IV from day 1 to day 4) every 3 weeks or Carboplatin (AUC 5 IV on day 1) + 5-FU (1000 mg/m^2 continuous IV from day 1 to day 4) every 3 weeks.
Period: Overall Study
Arm/Group | Cetuximab Plus Chemotherapy | Chemotherapy Alone
Started | 222 (Intention To Treat population, treatment group as randomized) | 220 (Intention To Treat population, treatment group as randomized)
Completed | 215 | 219
Not Completed | 7 | 1
Not completed — investigational study phase ongoing | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetuximab Plus Chemotherapy | Chemotherapy Alone | Total
Number analyzed (Participants) | 222 | 220 | 442
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 183 | 182 | 365
  >=65 years | 39 | 38 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (8.0) | 56.7 (8.7) | 56.9 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 18 | 43
  Male | 197 | 202 | 399
Region of Enrollment [Number; unit: participants]
  Portugal | 3 | 6 | 9
  Slovakia | 3 | 1 | 4
  Spain | 38 | 41 | 79
  Ukraine | 18 | 16 | 34
  Austria | 4 | 10 | 14
  Russian Federation | 9 | 7 | 16
  United Kingdom | 4 | 5 | 9
  Switzerland | 4 | 4 | 8
  Italy | 14 | 12 | 26
  France | 45 | 31 | 76
  Czech Republic | 4 | 5 | 9
  Hungary | 19 | 24 | 43
  Belgium | 14 | 16 | 30
  Poland | 18 | 18 | 36
  Germany | 18 | 14 | 32
  Netherlands | 4 | 6 | 10
  Sweden | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Time (OS)
Description: Time from randomization to death. Patients without event are censored at the last date known to be alive or at the clinical cut-off date, whatever is earlier.
Time Frame: time from randomization to death or last day known to be alive, reported between day of first patient randomised, 21 Dec 2004, until cut-off date 12 Mar 2007
Population: Primary analysis on Intent to Treat (ITT) population (allocation to treatment groups as randomized).
  Analysis performed after the required number of 340 deaths had been reported (expected effect: 36% increase in median survival time, power = 80%, alpha=5% (two-sided)). The Clinical cut-off date was 12 Mar 2007.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 222 | 220
months | 10.1 [8.6 to 11.2] | 7.4 [6.4 to 8.3]
Statistical Analysis 1: Comparison: Cetuximab Plus Chemotherapy vs Chemotherapy Alone; The primary analysis tested the equality of OS between treatment groups applying a 2-sided stratified log-rank test (α=5%), taking into account the strata used for randomization (previous chemotherapy (CTX) [no vs. yes] and Karnofsky Performance Status (KPS) [<80 vs. ≥80]). Median overall survival was estimated using the Kaplan-Meier method. The Hazard Ratio (HR) of cetuximab + CTX over CTX alone was calculated using the Cox proportional hazards model stratified by randomization strata; Test type: Superiority or Other; p = 0.036, Stratified Log Rank; Hazard Ratio (HR) = 0.797, 95% CI 2-sided [0.644 to 0.986]

2. Secondary Outcome: Progression-free Survival Time (PFS)
Description: Duration from randomization until radiological progression according to investigator (based on modified World Health Organisation (WHO) criteria) or death due to any cause.
  Only deaths within 60 days of last tumor assessment are considered. Patients without event are censored on the date of last tumor assessment.
Time Frame: time from randomization to disease progression, death or last tumor assessment, reported between day of first patient randomised, 21 Dec 2004, until cut-off date 12 Mar 2007
Population: Analysis on ITT population (allocation to treatment groups as randomized). Analysis performed at clinical cut off date, determined by primary endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 222 | 220
months | 5.6 [5.0 to 6.0] | 3.3 [2.9 to 4.3]
Statistical Analysis 1: Comparison: Cetuximab Plus Chemotherapy vs Chemotherapy Alone; To test the equality of PFS between treatment groups, a two-sided stratified log-rank test (α=5%)was used, taking into account strata used for randomization (previous CTX [yes/no] and KPS [<80 vs. ≥80]). Median PFS time was estimated using the Kaplan-Meier method. The HR of cetuximab + CTX over CTX alone was calculated using the Cox proportional hazards model stratified by randomization strata; Test type: Superiority or Other; p < 0.0001, Stratified Log Rank; Hazard Ratio (HR) = 0.538, 95% CI 2-sided [0.431 to 0.672]

3. Secondary Outcome: Best Overall Response
Description: The best overall response rate is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response as the best overall response according to radiological assessments according to investigator (based on modified WHO criteria).
Time Frame: evaluations were performed every 6 weeks until progression, reported between day of first patient randomised, 21 Dec 2004, until cut-off date 12 Mar 2007
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 222 | 220
percentage of participants | 35.6 [29.3 to 42.3] | 19.5 [14.5 to 25.4]
Statistical Analysis 1: Comparison: Cetuximab Plus Chemotherapy vs Chemotherapy Alone; A Cochran-Mantel-Haenszel (CMH) test was performed using the randomization strata previous CTX (no vs. yes) and KPS (<80 vs. ≥80). Treatment group comparisons were performed two-sided with α=5%; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.326, 95% CI 2-sided [1.504 to 3.600]

4. Secondary Outcome: Disease Control
Description: The disease control rate is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response + Stable Disease as best overall response according to radiological assessments according to investigator (based on modified WHO criteria).
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 222 | 220
percentage of participants | 81.1 [75.3 to 86.0] | 60.0 [53.2 to 66.5]
Statistical Analysis 1: Comparison: Cetuximab Plus Chemotherapy vs Chemotherapy Alone; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.881, 95% CI 2-sided [1.870 to 4.441]

5. Secondary Outcome: Time to Treatment Failure
Description: Time from randomization to date of the first occurrence of; progression, discontinuation of treatment due to progression or adverse event, start of new anticancer therapy, withdrawal of consent, or death (within 60 days of last tumor assessment).
  Patients without event are censored on the date of last tumor assessment.
Time Frame: Time from randomization to treatment failure or last tumor assessment, reported between day of first patient randomised, 21 Dec 2004, until cut-off date 12 Mar 2007
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 222 | 220
months | 4.8 [4.0 to 5.6] | 3.0 [2.8 to 3.4]
Statistical Analysis 1: Comparison: Cetuximab Plus Chemotherapy vs Chemotherapy Alone; Treatment groups were compared applying a two-sided stratified log-rank test (α=5%), taking into account strata used for randomization (previous CTX [yes/no] and KPS [<80 vs. ≥80]). Median time to treatment failure was estimated using the Kaplan-Meier method. The HR of cetuximab + CTX over CTX alone was calculated using the Cox proportional hazards model stratified by randomization strata; Test type: Superiority or Other; p < 0.0001, Stratified Log Rank; Hazard Ratio (HR) = 0.593, 95% CI 2-sided [0.484 to 0.727]

6. Secondary Outcome: Duration of Response
Description: Time from first assessment of Complete Response or Partial Response to disease progression or death (within 60 days of last tumor assessment).
  Patients without event are censored on the date of last tumor assessment. Tumor assessments based on modified WHO criteria.
Time Frame: time from first assessment of Complete Response or Partial Response to disease progression, death or last tumor assessment, reported between day of first patient randomised, 21 Dec 2004, until cut-off date 12 Mar 2007
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 222 | 220
months | 5.6 [4.7 to 6.0] | 4.7 [3.5 to 5.9]
Statistical Analysis 1: Comparison: Cetuximab Plus Chemotherapy vs Chemotherapy Alone; To test the equality of duration of response between treatment groups, the two-sided stratified log-rank test (α=5%) was used taking strata used for randomization into account (previous CTX [no vs. yes] and KPS [<80 vs. ≥80]). Median duration of response was estimated using the Kaplan-Meier method. The HR of cetuximab + CTX over CTX alone was calculated using the Cox proportional hazards model stratified by randomization strata; Test type: Superiority or Other; p = 0.21, Stratified Log Rank; Hazard Ratio (HR) = 0.762, 95% CI 2-sided [0.497 to 1.168]

7. Secondary Outcome: Quality of Life (QOL) Assessment European Organisation for the Research and Treatment of Cancer (EORTC) QLQ-C30 Global Health Status
Description: Mean global health status scores (EORTC QLQ-C30) against time for each treatment group. Scores were derived from mutually exclusive sets of items, with scale scores ranging from 0 to 100 after a linear transformation. Higher scores indicate a better QoL.
Time Frame: at baseline, day 1 of cycle 3, first 6-weekly evaluation following completion of chemotherapy, 6 & 12 months after randomization, reported between day of first patient randomised, 21 Dec 2004,until cut-off date, 12 Mar 2007
Population: Of 361 ITT subjects from countries with EORTC QLQ-C30 available, 291 completed ≥1 evaluable questionnaire. Only time points where ≥ 20% of patients completing a baseline questionnaire remained in the population were analysed. Numbers at each timepoint were (cetuximab+chemotherapy/chemotherapy alone): Baseline: 121/106; Cycle3:87/67; Month6:48/22
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Cetuximab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 152 | 139
scores on a scale
  At baseline | 50.74 (3.519) | 45.15 (3.745)
  At cycle 3 | 52.68 (3.724) | 45.48 (4.153)
  Month 6 | 55.30 (4.282) | 42.49 (5.959)

8. Secondary Outcome: Quality of Life Assessment (EORTC QLQ-C30) Social Functioning
Description: Mean social functioning scores (EORTC QLQ-C30) against time for each treatment group. Scores were derived from mutually exclusive sets of items, with scale scores ranging from 0 to 100 after a linear transformation. Higher scores indicate a higher level of social functioning.
Time Frame: as for outcome 7
Population: Of 361 ITT subjects from countries with EORTC QLQ-C30 available, 291 completed ≥1 evaluable questionnaire. Only time points where ≥ 20% of patients completing a baseline questionnaire remained in the population were analysed. Numbers at each timepoint were (cetuximab +chemotherapy/chemotherapy alone): Baseline:123/109; Cycle3:87/69; Month6:48/23
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Cetuximab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 152 | 139
scores on a scale
  At baseline | 62.14 (4.459) | 62.05 (4.730)
  At cycle 3 | 64.64 (4.663) | 60.67 (5.176)
  Month 6 | 61.27 (5.347) | 65.72 (7.122)

9. Secondary Outcome: Safety - Number of Patients Experiencing Any Adverse Event
Description: Please refer to Adverse Events section for further details
Time Frame: time from first dose up to 30 after last dose of study treatment, reported between day of first dose of study treatment, 22 Dec 2004, until cut-off date 12 Mar 2007
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Cetuximab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 219 | 215
participants | 218 | 208

ADVERSE EVENTS:
Time Frame: Time from first dose up to 30 days after the last dose of study treatment.
Description: Treatment-emergent adverse events were defined as those with onset occurring at or after the first dosing day of study medication and up to 30 days after the last administration of any study drug or the clinical cut-off date.
Arm/Group | Cetuximab Plus Chemotherapy | Chemotherapy Alone
Serious Adverse Events (participants affected / at risk) | 110/219 | 102/215
Other Adverse Events (participants affected / at risk) | 214/219 | 198/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab Plus Chemotherapy (N=219) | Chemotherapy Alone (N=215)
Anaemia (Blood and lymphatic system disorders) | 5 | 10
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 9
Haemolysis (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 5
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 10
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 6
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 1
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 2
Cardiac failure (Cardiac disorders) | 2 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 2 | 0
Coronary artery thrombosis (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 0 | 1
Keratitis (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Aphagia (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 0
Stress ulcer (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 5 | 4
Asthenia (General disorders) | 2 | 1
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Death (General disorders) | 1 | 1
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 4 | 2
General physical health deterioration (General disorders) | 5 | 2
Hyperthermia (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 5 | 6
Multi-organ failure (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Performance status decreased (General disorders) | 2 | 4
Pyrexia (General disorders) | 2 | 7
Sudden death (General disorders) | 2 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 4 | 0
Abscess neck (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 1
Catheter related infection (Infections and infestations) | 2 | 0
Catheter sepsis (Infections and infestations) | 1 | 0
Central line infection (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Lymph gland infection (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 10 | 4
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Pyothorax (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 2
Salmonella sepsis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 6 | 1
Septic shock (Infections and infestations) | 3 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Thrombophlebitis septic (Infections and infestations) | 0 | 1
Feeding tube complication (Injury, poisoning and procedural complications) | 1 | 0
Gastrostomy failure (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 1
Blood creatinine increased (Investigations) | 1 | 1
Creatinine renal clearance decreased (Investigations) | 1 | 0
Haemoglobin (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 4
Neurological examination abnormal (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Urine electrolytes decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 3
Anorexia (Metabolism and nutrition disorders) | 3 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 9 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 7
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain oedema (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 1
Coma (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 2 | 3
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 0
Intracranial hypotension (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 3
Confusional state (Psychiatric disorders) | 1 | 3
Suicide attempt (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 2
Renal failure acute (Renal and urinary disorders) | 3 | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 11
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 0
Gastrostomy tube insertion (Surgical and medical procedures) | 1 | 0
Medical device removal (Surgical and medical procedures) | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
Haemorrhage (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 2
Ischaemia (Vascular disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 1
Thrombosis (Vascular disorders) | 2 | 1
Wound haemorrhage (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab Plus Chemotherapy (N=219) | Chemotherapy Alone (N=215)
Anaemia (Blood and lymphatic system disorders) | 92 | 111
Neutropenia (Blood and lymphatic system disorders) | 83 | 77
Thrombocytopenia (Blood and lymphatic system disorders) | 46 | 48
Leukopenia (Blood and lymphatic system disorders) | 41 | 32
Lymphopenia (Blood and lymphatic system disorders) | 16 | 13
Conjunctivitis (Eye disorders) | 21 | 0
Nausea (Gastrointestinal disorders) | 119 | 100
Vomiting (Gastrointestinal disorders) | 84 | 79
Diarrhoea (Gastrointestinal disorders) | 56 | 33
Constipation (Gastrointestinal disorders) | 48 | 43
Stomatitis (Gastrointestinal disorders) | 31 | 28
Dysphagia (Gastrointestinal disorders) | 21 | 19
Dyspepsia (Gastrointestinal disorders) | 15 | 7
Abdominal pain upper (Gastrointestinal disorders) | 13 | 7
Asthenia (General disorders) | 56 | 47
Mucosal inflammation (General disorders) | 50 | 38
Fatigue (General disorders) | 49 | 44
Pyrexia (General disorders) | 48 | 23
General physical health deterioration (General disorders) | 11 | 2
Paronychia (Infections and infestations) | 19 | 0
Weight decreased (Investigations) | 41 | 30
Platelet count decreased (Investigations) | 13 | 7
Blood creatinine increased (Investigations) | 11 | 13
Haemoglobin decreased (Investigations) | 9 | 11
Anorexia (Metabolism and nutrition disorders) | 54 | 31
Hypocalcaemia (Metabolism and nutrition disorders) | 26 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 25 | 15
Hypomagnesaemia (Metabolism and nutrition disorders) | 22 | 11
Hyponatraemia (Metabolism and nutrition disorders) | 12 | 17
Hyperkalaemia (Metabolism and nutrition disorders) | 12 | 11
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 | 19
Headache (Nervous system disorders) | 20 | 15
Peripheral sensory neuropathy (Nervous system disorders) | 14 | 8
Dizziness (Nervous system disorders) | 10 | 11
Insomnia (Nervous system disorders) | 20 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 19
Productive cough (Respiratory, thoracic and mediastinal disorders) | 12 | 12
Rash (Skin and subcutaneous tissue disorders) | 61 | 4
Acne (Skin and subcutaneous tissue disorders) | 48 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 32 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 30 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 27 | 15
Pruritus (Skin and subcutaneous tissue disorders) | 18 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 17 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 13 | 0
Hypertension (Vascular disorders) | 15 | 10
Hypotension (Vascular disorders) | 14 | 9
Phlebitis (Vascular disorders) | 11 | 5

LIMITATIONS AND CAVEATS:
Non-specific outcome measures 'Safety' & 'QOL assessments' were deleted from this entry in error.Replacement outcomes have been created. The 'Safety' outcome refers to adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other